CLINICAL TRIAL: NCT07379047
Title: A Multicenter, Open-label Clinical Study to Evaluate the Efficacy and Safety of NB003 in Patients With Advanced Gastrointestinal Stromal Tumors (GIST)
Acronym: GISTAR-1
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ningbo Newbay Technology Development Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NB003-04
Record Dates: First submitted 2026-01-23; First posted 2026-01-30 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: GIST - Gastrointestinal Stromal Tumor; Advanced
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — regorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- NB003 (Experimental): part1 treated arm
  Interventions: Drug: NB003
- Regorafenib (Active Comparator): 160 mg QD in 28-day cycles.
  Interventions: Drug: NB003; Drug: regorafenib
- NB003（part 2） (Experimental): part 2 single arm
  Interventions: Drug: NB003

INTERVENTIONS:
Drug: NB003 — 15 mg BID on a continuous schedule in 28-day cycles.
Drug: regorafenib — Regorafenib is an approved multi-kinase inhibitor administered orally at a dose of 160 mg once daily (QD).
  Arms: Regorafenib

SUMMARY:
NB003-04 is a phase II/III, multicenter, open-label clinical study designed to evaluate the efficacy, safety, and pharmacokinetic (PK) profile of NB003 in patients with gastrointestinal stromal tumors aged 18 years and above (or the legal adult age of consent per local regulations, whichever is older). Participants who are eligible for this study are those who have experienced disease progression or documented intolerance following treatment with either imatinib and sunitinib or following treatment with imatinib.

This study consists of two parts. Part 1 (hereinafter referred to as Part 1) compares the efficacy of NB003 versus regorafenib in patients who need a third-line therapy for GIST who have failed sequential therapy with imatinib and sunitinib. Part 2 (hereinafter referred to as Part 2) evaluates the efficacy of NB003 in patients who need a second-line therapy for GIST who have failed treatment with imatinib.

ELIGIBILITY:
Inclusion Criteria:

1. Participants are >=18 years of age (or the legal adult age as per local regulations, whichever is older) at the time of signing the ICF.
2. Participants, or legally authorized representatives permitted by local regulations, provide written informed consent for participation in the study.
3. Participants who have histologically confirmed locally advanced, unresectable, or metastatic GIST.

   1. Part 1: Patients who have failed prior treatment with imatinib (including adjuvant therapy) and sunitinib for GIST due to disease progression or intolerance. Participants should also have no prior use of other TKI drugs.
   2. Part 2: Patients who have failed prior treatment with imatinib (including adjuvant therapy) for GIST due to disease progression or intolerance. Participants should also have no prior use of other TKI drugs.
4. Participants with confirmed KIT gene mutation based on local or central laboratory molecular pathology reports. Mutation status must be determined using tissue-based PCR or DNA sequencing methods. The report should include results on the presence or absence of KIT exon 9/11/17 mutations for randomization stratification in Part 1 and efficacy-related analyses throughout the study. The molecular pathology report indicating KIT mutation status shall be submitted to the medical monitor for review during the screening period. If a local molecular pathology report is unavailable or provides insufficient information, archived tumor tissue samples or fresh biopsy samples must be provided for central laboratory confirmation of mutation status prior to enrollment.
5. Participants with at least one measurable lesion according to mRECIST.
6. Participants with an ECOG PS of 0 to 1.
7. Tumor sample requirement: Archival tumor samples in the form of formalin-fixed paraffin-embedded (FFPE) tissue sections or FFPE blocks obtained prior to enrollment, or tissue samples from a tumor biopsy (excisional, core needle, or fine-needle aspiration).
8. Participants with an expected life expectancy of >=12 weeks.
9. Participants shall have adequate organ and bone marrow function. Transfusions and/or treatment with erythropoietin and/or granulocyte colony stimulating factor/granulocyte macrophage colony stimulating factor (G-CSF/GM-CSF) are not permitted within 14 days prior to the screening laboratory blood draw under any circumstances. The criteria are defined as follows:

   * Hemoglobin >=9 g/dL (5.59 mmol/L).
   * Absolute neutrophil count (ANC) >=1.5 x 10^9/L (1500/mm^3).
   * Platelet count >=100 x 10^9/L (100,000/mm^3).
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <= 2.5 x upper limit of normal (ULN) (for participants without liver metastases); AST and ALT <= 5 x ULN (for participants with liver metastases).
   * Total bilirubin <=1.5 x ULN. Participants with a confirmed diagnosis of Gilbert's syndrome (persistent or recurrent unconjugated hyperbilirubinemia in the absence of hemolysis or hepatic pathology) may be enrolled if total bilirubin <=3 x ULN.
   * Creatinine clearance >=60 mL/min as calculated by the Cockcroft-Gault formula or 24-hour urine collection.
   * International normalized ratio (INR) or prothrombin time (PT) and activated partial thromboplastin time (aPTT) <=1.5 x ULN; however, if a participant is receiving anticoagulant therapy, PT or aPTT within the therapeutic range of the anticoagulant is acceptable.
10. Male participants: Male participants must agree to use contraception as detailed in Appendix 9 during the treatment period and for at least 6 months after the last dose of study treatment and refrain from donating sperm during this period.
11. Female participants: A female participant is eligible to participate if she is not pregnant, not breastfeeding, and at least one of the following conditions applies:

    i) She is not a woman of childbearing potential (WOCBP) as defined in the Appendix 9; or ii) She is a WOCBP and agrees to follow the contraceptive guidance outlined in the Appendix 9 during the treatment period and for at least 6 months after the last dose of study treatment.
12. WOCBP must have a negative serum pregnancy test result during screening within 14 days prior to enrollment.

Exclusion Criteria:

1. Part 1: Participants who have received prior treatment with NB003 or regorafenib. Part 2: Participants who have received prior treatment with NB003 or sunitinib.
2. Participants who have received any systemic anti-tumor therapy within 7 days prior to enrollment.
3. Participants who have undergone major surgery (excluding vascular access placement, tumor biopsy, and feeding tube placement) or major palliative interventions (such as transarterial chemoembolization) within 4 weeks prior to enrollment.
4. Participants who have received radiation therapy to >30% of the bone marrow or extensive radiation therapy within 4 weeks prior to enrollment.
5. Active infection, including active hepatitis B [defined as detectable HBV-DNA by local laboratory. Participants who are HBsAg positive or HBcAb positive at screening should have HBV-DNA tested] and active hepatitis C [defined as detectable HCV-RNA by local laboratory. Participants who are HCV antibody positive at screening should have HCV-RNA tested].
6. Any of the following cardiac-related criteria:

   * Uncontrolled persistent (>4 weeks) hypertension (>140/90 mmHg).
   * New York Heart Association (NYHA) Class (Appendix 11) III and IV heart disease, active ischemia, or other uncontrolled cardiac conditions such as angina.
   * QTc interval Corrected QT interval using Fridericia's formula (QTcF) >=470 ms (based on 3 ECG results) or history of long QT syndrome.
   * Resting ECG showing any clinically significant abnormalities in rhythm, conduction, or morphology (e.g., complete left bundle branch block, atrioventricular block third degree, atrioventricular block second degree, PR interval >250 ms).
   * Left ventricular ejection fraction (LVEF) <50%.
7. Any unresolved prior treatment toxicity greater than CTCAE Grade 1 at the start of study treatment, with the exception of alopecia, hemoglobin (see Inclusion Criterion #10), Grade 2 hypothyroidism stable on hormone replacement therapy, and Grade 2 pre-existing treatment-related neuropathy.
8. Participants who have experienced a National Cancer Institute Common Terminology Criteria for Adverse Events version 5.0 Grade 3 or higher bleeding event within 4 weeks prior to enrollment.
9. Participants who have experienced an arterial thrombotic or embolic event (e.g., cerebrovascular accident, including transient ischemic attack) within 6 months prior to enrollment, or a venous thrombotic event (including pulmonary embolism or deep vein thrombosis) within 3 months prior to enrollment.
10. Participants who have experienced a seizure for any reason within 6 months prior to enrollment.
11. Participants with known bleeding disorders or risk of intracranial hemorrhage (e.g., unexcised or unrepaired cerebral aneurysm, cerebrovascular malformation), or history of intracranial hemorrhage within 1 year prior to randomization.
12. Participants with unhealed wounds, active ulceration, gastrointestinal perforation, or fracture within 3 months prior to enrollment.
13. Participants with brain metastases.
14. History of pancreatitis with prior tyrosine kinase inhibitors use, or current evidence of mild to moderate pancreatitis.
15. Refractory nausea and vomiting, chronic gastrointestinal disease, inability to swallow the formulation, or significant bowel resection that may affect adequate absorption of NB003 and regorafenib.
16. Any other clinically significant comorbidity, such as uncontrolled lung disorder, active infection, uncontrolled pericardial effusion, uncontrolled pleural effusion, or any other condition that, in the investigator's judgment, may affect protocol compliance, interfere with interpretation of study results, or increase participant safety risk.
17. Participants judged by the investigator to be unwilling or unable (including incompetence) to comply with study procedures, restrictions, and requirements.
18. Participants currently using (or unable to discontinue at least 2 weeks prior to enrollment) drugs or herbal supplements known to be strong inhibitors or inducers of CYP3A4, and other prohibited concomitant medications (Appendix 3).
19. History of hypersensitivity to the active or inactive ingredients of NB003, regorafenib, or drugs with similar chemical structure or class to NB003 or regorafenib.
20. History of other primary neoplasm malignant diagnosed or requiring treatment within 3 years prior to enrollment. The following prior malignancies are not exclusion criteria: completely resected basal cell and squamous cell skin cancers, cured localized prostate cancer, cured superficial or non-muscle invasive bladder cancer, and completely resected carcinoma in situ of any site.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 255 (Estimated)
Dates: Start 2026-04-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2028-09-01 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival (PFS) | From randomization until database cut-off, approximately 28 months
  for part 1
Objective response rate (ORR) | approximately 24 months since the first subject enrolled
  for part 2

SECONDARY OUTCOMES:
Objective response rate (ORR) | From randomization until database cut-off, approximately 28 months
  for part 1
Progression-free survival (PFS) | approximately 24 months since the first subject enrolled
  for part 2
Duration of Response(DOR) | approximately 24 months since the first subject enrolled
  for part 2
Duration of Response(DOR) | approximately 28 months since the first subject enrolled
  for part 1
Overall Survival(OS) | approximately 24-36 months
  for part 1
Disease Control Rate (DCR) | Approximately 28 months since first subject enrolled
  for part 1
Overall Survival(OS) | approximately 24-36 months
  for part 2
Disease Control Rate (DCR) | Approximately 24 months since first subject enrolled
  for part 2

CONTACTS AND LOCATIONS:
Locations (9):
- China (9):
  - The Second Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guandong
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Xiangya Hospital, Central South University, Changsha, Huanan
  - The Affiliated Hospital of Qingdao University, Qingdao, Shandong
  - Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - The First Affiliated Hospital of Zhejiang University School of Medicine, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided